CLINICAL TRIAL: NCT06991127
Title: Pre-market Multicentric Cross-sectional Clinical Investigation of MAIA Microperimeter Device: Mesopic Normative Database Collection
Brief Title: Clinical Investigation of MAIA Microperimeter Device: Mesopic Normative Database Collection
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Centervue SpA (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: MAIA_003_MNDB
Record Dates: First submitted 2025-05-19; First posted 2025-05-25 (Actual); Last update posted 2025-05-25 (Actual); Status verified 2025-04

CONDITIONS: Healthy Eyes

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (1):
- Main Arm (Experimental): *) one microperimetric examination with MAIA
  Interventions: Device: MAIA

INTERVENTIONS:
Device: MAIA — MAIA is an automatic microperimeter with fundus imaging capabilities that measures retinal sensitivity, fixation stability and locus of fixation, and allows the acquisition of confocal images of the retina, thanks to its confocal scanning imaging system which uses infrared and visible light.

SUMMARY:
The purpose of this pre-market, multicentric cross-sectional study is to create a mesopic Normative Database for a new version of the MAIA device. Moreover, the study aims to evaluate MAIA safety and adverse events. These purposes will be achieved by collecting data of healthy subjects, who will undergo microperimetric examinations with the MAIA device during one single visit.

ELIGIBILITY:
Inclusion Criteria:

* Age: ≥18 years old;
* Best Corrected Visual Acuity (BCVA): ≥ 0.8 Decimal (≥ 20/25 ft, ≤ +0.1 logMAR) at least in the study eye;
* Equivalent spherical refraction between the range ≥ -6D and ≤ +6D; astigmatism within 2D (≤ 2D) at least in the study eye;
* Intraocular Pressure (IOP) ≤ 21 mmHg in both eyes (Goldmann applanation tonometer);
* Clinically normal appearance of the optic nerve head according to clinical judgement (no evidence of excavation, rim thinning, notching, disc hemorrhages, RNFL thinning) in both eyes. This is examined with Spectralis or Solix OCT;
* Clinically normal appearance of the macula according to clinical judgement, in both eyes. This is examined with Spectralis or Solix OCT;
* No ocular pathologies, trauma, surgeries (apart from uncomplicated cataract surgery or peripheral laser retinopexy performed at least 6 months before enrollment) in both eyes;
* Absence of pathologies that can affect visual field in both eyes;
* No use of drugs interfering with the correct execution of perimetry.

Exclusion Criteria:

* Glaucoma or glaucoma suspect diagnosis in either eye;
* Presence or history of ocular hypertension (IOP ≥ 22 mmHg) in either eye;
* Presence or history of disc hemorrhage in either eye;
* Presence of amblyopia in either eye;
* Nystagmus or poor fixation in either eye;
* Previous laser or any ocular surgery, including uncomplicated cataract surgery performed within 6 months before enrollment in both eyes;
* Any active infection of anterior or posterior segments in the study eye;
* Subjects with significant ocular media opacities preventing acquisition of acceptable infrared (IR) fundus image quality in the study eye;
* Evidence of diabetic retinopathy, diabetic macular edema, or other retinal disease in either eye;
* Use of any drug that can interfere with the correct execution of MP or that would produce visual field loss;
* Unable to tolerate ophthalmic imaging;
* Claustrophobia;
* Inability to provide informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 380 (Estimated)
Dates: Start 2025-04-23 (Actual); Primary Completion 2026-05-01 (Estimated); Study Completion 2026-06-01 (Estimated)

PRIMARY OUTCOMES:
To determine the reference normative values of retinal sensitivity for MAIA | 1 day
  The reference normative values will be determined by using a linear regression model for Mean Sensitivity (MS) as a function of age. The 5th and 10th percentile values will be derived for each age, and will serve as age-adjusted normative data against which compare the MS computed during each test with MAIA

SECONDARY OUTCOMES:
To assess the avoidance of Serious Adverse Device Effects with MAIA | through study completion (expected duration: 10 months)
  During the clinical investigation, adverse events will be documented, investigated and reported according to the provisions of applicable reporting guidelines, following their criteria and timelines.

CONTACTS AND LOCATIONS:
Overall Officials: Maximilian Pfau, PD Dr. med., Study Chair — Universitätsspital Basel, Augenklinik
Locations (3):
- The Eye Care Institute, Fort Lauderdale, Florida, United States
- UWA Eye Health Centre of Western Australia, Perth, Western Australia, Australia
- Universitätsspital Basel, Augenklinik, Basel, Switzerland, Switzerland

IPD SHARING:
Plan to Share IPD: No